CLINICAL TRIAL: NCT04450277
Title: Delivery of Protocolised Emergency Surgical Care During COVID-19 Pandemic Based on Case Series
Brief Title: Delivery of Protocolised Emergency Surgical Care During COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Khoo Teck Puat Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/00660
Record Dates: First submitted 2020-06-25; First posted 2020-06-29 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: COVID-19; Emergency Surgery
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Emergency surgery — Emergency surgery vs conservative management

SUMMARY:
Emergency general surgical care during the COVID-19 pandemic presents a unique set of considerations and challenges. Patients presenting with acute surgical conditions and concomitant COVID-19 infection have higher risk of mortality and morbidity. The investigators present their experience with COVID-19 positive patients presenting with acute surgical conditions and reviewed the implementation of a protocolized pathway to mitigate the impact of COVID-19 infection.

DETAILED DESCRIPTION:
All COVID-19 positive patients who presented to the acute general surgical service over a 2-month period were identified. Patient data including demographics, surgical diagnosis, mortality, morbidity and hospital length of stay was collected. Based on the investigators' early experience from the first patient, the investigators designed a protocolized institutional pathway which incorporated the risk of COVID-19 infection and urgency of operation.

ELIGIBILITY:
Inclusion Criteria:

* All patients with emergency surgical conditions and tested positive for COVID-19 infection

Exclusion Criteria:

* Nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A propsective review was performed of all patients with laboratory-confirmed COVID-19 infection who presented with acute general surgical conditions to Khoo Teck Puat Hospital (KTPH), in the period of 1st April 2020 to 31st May 2020. KTPH is a 795-bed regional general hospital in Singapore that serves approximately half a million people in the northern part of the city state. A confirmed case of COVID-19 was defined by a positive result on a reverse-transcriptase-polymerase-chain-reaction (RT-PCR) assay of a specimen collected on a nasopharyngeal swab. Patients underwent testing on admission if identified as high risk as per national guidelines, or upon developing respiratory symptoms during inpatient stay.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Surgical morbidity in patients with COVID-19 infection and general surgical conditions | Follow up 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Khoo Teck Puat Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data due to personal data protection act